CLINICAL TRIAL: NCT04051203
Title: Ultrasound Guided Platelet Rich Plasma Injections for Post Traumatic Greater Occipital Neuralgia: A Randomized Controlled Pilot Study
Brief Title: Ultrasound Guided Platelet Rich Plasma Injections for Post Traumatic Greater Occipital Neuralgia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: REB18-1368
Record Dates: First submitted 2019-07-23; First posted 2019-08-09 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2023-10

CONDITIONS: Occipital Neuralgia; Headache
Keywords: GON; greater occipital neuralgia; post traumatic headache; post concussive headache
MeSH Terms: conditions — Headache; Post-Traumatic Headache | interventions — Methylprednisolone Acetate; Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, participants are randomly assigned to one of three groups; an autologous PRP injection, a steroid injection, or normal saline.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All members of the study will be blinded (participants and healthcare practioners) except for the study coordinator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Autologous Platelet Rich Plasma Injection (Experimental): PRP contains high concentrations of platelets, growth factors, and anti-inflammatory molecules.
  Interventions: Biological: Autologous Platelet Rich Plasma Injection
- Standard Treatment (Active Comparator): Steroid and anesthetic injection: the clinical standard.
  Interventions: Drug: Depo-Medrol and lidocaine
- Normal Saline (Placebo Comparator): Placebo injection, with no known treatment effects.
  Interventions: Other: Normal Saline

INTERVENTIONS:
Biological: Autologous Platelet Rich Plasma Injection — 60mL of blood will be drawn from the antecubital vein and processed via centrifugation. Samples will be centrifuged as per manufacturer instructions, yielding 5mL of PRP.
  Arms: Autologous Platelet Rich Plasma Injection
Drug: Depo-Medrol and lidocaine — Steroid injections will be prepared to include 20mg Depo-Medrol and 2mL 2% lidocaine.
  Arms: Standard Treatment
Other: Normal Saline — 2mL normal saline.
  Arms: Normal Saline

SUMMARY:
This study is a randomized controlled trial, assessing the effect of a single platelet rich plasma (PRP) injection in post traumatic (concussive) greater occipital neuralgia. This study will compare the effects of a single PRP injection to injection with steroid and anesthetic. There will also be a third arm to the study, in which patients will receive an injection with normal saline. This study will assess the severity and frequency of headache symptoms before and after receiving the injection.

DETAILED DESCRIPTION:
Each year, an estimated 69 million people suffer from traumatic brain injury/concussion worldwide. In most patients with concussion, symptoms improve within 3 months. However, in some persons, symptoms persist. The cause(s) of post-traumatic headache are not entirely clear, which limits treatment options. Sometimes, these headaches are caused by irritation to the greater occipital nerve, and pain originating from this area is called "greater occipital neuralgia". These headaches are often treated with steroid injections to the affected nerve. However, the effect of the injection is usually short lasting and may not provide adequate pain relief.

Therefore, other methods of treatment have been sought out. Platelet Rich Plasma (PRP) is an emerging biologic treatment. PRP contains high concentrations of platelets, growth factors, and anti-inflammatory molecules. PRP acts to reduce inflammation and encourage tissue repair at the site of injection. PRP is created by collecting a person's own blood, centrifuging it, and extracting the platelet-rich layer of plasma. This platelet rich mixture is then re-injected into the affected area. PRP is used as a safe and effective treatment in many fields, and is most commonly used in arthritis. PRP has recently been studied as a potential treatment for peripheral nerve disorders, such as carpal tunnel syndrome.

Post-injection, a daily headache diary provided via mobile application (Secure RedCap) available in iPhone or android device will be provided to record daily records of numeric pain rating scale, headache frequency and medication-use.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be males or females at least 18 years of age who suffer from post-traumatic headaches secondary to GON. Patients must fulfill the ICHD-3 criteria in establishing a diagnosis of GON. This diagnosis will be established by an experienced Physiatrist with extensive experience in headache and related disorders. To meet this criteria, patients must have experienced previous successful temporary relief with local anesthetic or steroid injection surrounding the GON in the past, but have not received local steroid injection within past 3 months. Pre-treatment numerical pain rating scale for daily headache intensity must be ≥4/10, with a headache frequency ≥10 days/month. Possible secondary causes of ON must be ruled out with reasonable level of investigation prior to enrollment.

Exclusion Criteria:

* Inability to provide informed consent; history of surgery in the occipital region; unstable psychiatric or medical condition; rheumatologic or inflammatory disorders; widespread neurologic disorders (eg. MS); coagulopathy; immunosuppression; active cancer; herpes zoster infection in last 6 months; pregnancy; steroid or other local GON or LON infiltration in past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of platelet-rich plasma for patients with post-traumatic greater occipital neuralgia | Screening, pre-injection to 3-months post injection
  The feasibility will be determined based on recruitment (greater than 30% of those screened eligible), attendance (70% intervention appointment attendance), retention (70% complete study protocol), and the acceptability of the protocol
Evaluate the safety profile of platelet-rich plasma for the treatment of post-traumatic greater occipital neuralgia | from immediately post-injection to 3-months, daily recording
  Safety will be determined based on adverse reactions monitored through daily headache diary reporting and communication with the study team

SECONDARY OUTCOMES:
Change in headache severity as measured by the Numerical Pain Raiting Scale (NPRS) | Pre-injection to 3 months post injection, daily recording.
  This will be measured as a greater than a 2-point decrease on the NPRS at 3 months post-injection in the PRP group as compared to steroid and saline groups.
Change in headache frequency (days per month with headache). | Pre-injection to 3 months post injection, daily recording.
  Using daily headache diaries, headache frequency will be collected.
Headache Impact Test-6 | Pre-injection, 1 month, and 3 month time points.
  A valid and reliable 6-item questionnaire for assessment of the impact of headaches across different diagnostic groups of headaches. The HIT-6 items measure the adverse impact of headache on social functioning, role functioning, vitality, cognitive functioning and psychological distress. The HIT-6 also measures the severity of headache pain.
Quality of Life in Following Brain Injury Questionnaire | Pre-injection, 1 month, and 3 month follow-ups.
  The QOLIBRI (Quality of Life after Brain Injury) is the first instrument specifically developed to assess health-related quality of life (HRQoL) of individuals after traumatic brain injury. The QOLIBRI is a comprehensive questionnaire with 37 items covering six dimensions of HRQoL after TBI. The questionnaire provides a profile of quality of life together with a total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Center, Main Floor Special Services, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
There is no plan, all participant data will be kept on a secured REDCap database.

REFERENCES:
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Hyder AA, Wunderlich CA, Puvanachandra P, Gururaj G, Kobusingye OC. The impact of traumatic brain injuries: a global perspective. NeuroRehabilitation. 2007;22(5):341-53. PMID 18162698
- [Background] Dewan MC, Rattani A, Gupta S, Baticulon RE, Hung YC, Punchak M, Agrawal A, Adeleye AO, Shrime MG, Rubiano AM, Rosenfeld JV, Park KB. Estimating the global incidence of traumatic brain injury. J Neurosurg. 2018 Apr 27;130(4):1080-1097. doi: 10.3171/2017.10.JNS17352. Print 2019 Apr 1. PMID 29701556
- [Background] Coronado VG, Xu L, Basavaraju SV, McGuire LC, Wald MM, Faul MD, Guzman BR, Hemphill JD; Centers for Disease Control and Prevention (CDC). Surveillance for traumatic brain injury-related deaths--United States, 1997-2007. MMWR Surveill Summ. 2011 May 6;60(5):1-32. PMID 21544045
- [Background] Ponsford JL, Downing MG, Olver J, Ponsford M, Acher R, Carty M, Spitz G. Longitudinal follow-up of patients with traumatic brain injury: outcome at two, five, and ten years post-injury. J Neurotrauma. 2014 Jan 1;31(1):64-77. doi: 10.1089/neu.2013.2997. PMID 23889321
- [Background] Lundin A, de Boussard C, Edman G, Borg J. Symptoms and disability until 3 months after mild TBI. Brain Inj. 2006 Jul;20(8):799-806. doi: 10.1080/02699050600744327. PMID 17060147
- [Background] Hoffman JM, Lucas S, Dikmen S, Braden CA, Brown AW, Brunner R, Diaz-Arrastia R, Walker WC, Watanabe TK, Bell KR. Natural history of headache after traumatic brain injury. J Neurotrauma. 2011 Sep;28(9):1719-25. doi: 10.1089/neu.2011.1914. Epub 2011 Aug 29. PMID 21732765
- [Background] Hammond SR, Danta G. Occipital neuralgia. Clin Exp Neurol. 1978;15:258-70. PMID 756019
- [Background] Dougherty C. Occipital neuralgia. Curr Pain Headache Rep. 2014 May;18(5):411. doi: 10.1007/s11916-014-0411-x. PMID 24737457
- [Background] Ward JB. Greater occipital nerve block. Semin Neurol. 2003 Mar;23(1):59-62. doi: 10.1055/s-2003-40752. PMID 12870106
- [Background] Anthony M. Headache and the greater occipital nerve. Clin Neurol Neurosurg. 1992;94(4):297-301. doi: 10.1016/0303-8467(92)90177-5. PMID 1335856
- [Background] Choi I, Jeon SR. Neuralgias of the Head: Occipital Neuralgia. J Korean Med Sci. 2016 Apr;31(4):479-88. doi: 10.3346/jkms.2016.31.4.479. Epub 2016 Mar 9. PMID 27051229
- [Background] Kuhn WF, Kuhn SC, Gilberstadt H. Occipital neuralgias: clinical recognition of a complicated headache. A case series and literature review. J Orofac Pain. 1997 Spring;11(2):158-65. PMID 10332322
- [Background] Laver L, Marom N, Dnyanesh L, Mei-Dan O, Espregueira-Mendes J, Gobbi A. PRP for Degenerative Cartilage Disease: A Systematic Review of Clinical Studies. Cartilage. 2017 Oct;8(4):341-364. doi: 10.1177/1947603516670709. Epub 2016 Sep 1. PMID 28317389
- [Background] Sampson S, Gerhardt M, Mandelbaum B. Platelet rich plasma injection grafts for musculoskeletal injuries: a review. Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):165-74. doi: 10.1007/s12178-008-9032-5. PMID 19468902
- [Background] Anitua E, Sanchez M, Orive G, Andia I. The potential impact of the preparation rich in growth factors (PRGF) in different medical fields. Biomaterials. 2007 Nov;28(31):4551-60. doi: 10.1016/j.biomaterials.2007.06.037. Epub 2007 Jul 30. PMID 17659771
- [Background] Park GY, Kwon DR. Platelet-rich plasma limits the nerve injury caused by 10% dextrose in the rabbit median nerve. Muscle Nerve. 2014 Jan;49(1):56-60. doi: 10.1002/mus.23863. Epub 2013 Sep 20. PMID 23558771
- [Background] Farrag TY, Lehar M, Verhaegen P, Carson KA, Byrne PJ. Effect of platelet rich plasma and fibrin sealant on facial nerve regeneration in a rat model. Laryngoscope. 2007 Jan;117(1):157-65. doi: 10.1097/01.mlg.0000249726.98801.77. PMID 17202946
- [Background] Sariguney Y, Yavuzer R, Elmas C, Yenicesu I, Bolay H, Atabay K. Effect of platelet-rich plasma on peripheral nerve regeneration. J Reconstr Microsurg. 2008 Apr;24(3):159-67. doi: 10.1055/s-2008-1076752. Epub 2008 Apr 30. PMID 18452111
- [Background] Ding XG, Li SW, Zheng XM, Hu LQ, Hu WL, Luo Y. The effect of platelet-rich plasma on cavernous nerve regeneration in a rat model. Asian J Androl. 2009 Mar;11(2):215-21. doi: 10.1038/aja.2008.37. Epub 2009 Jan 19. PMID 19151738
- [Background] Giannessi E, Coli A, Stornelli MR, Miragliotta V, Pirone A, Lenzi C, Burchielli S, Vozzi G, De Maria C, Giorgetti M. An autologously generated platelet-rich plasma suturable membrane may enhance peripheral nerve regeneration after neurorraphy in an acute injury model of sciatic nerve neurotmesis. J Reconstr Microsurg. 2014 Nov;30(9):617-26. doi: 10.1055/s-0034-1372483. Epub 2014 May 16. PMID 24838385
- [Background] Sanchez M, Anitua E, Delgado D, Prado R, Sanchez P, Fiz N, Guadilla J, Azofra J, Pompei O, Orive G, Ortega M, Yoshioka T, Padilla S. Ultrasound-guided plasma rich in growth factors injections and scaffolds hasten motor nerve functional recovery in an ovine model of nerve crush injury. J Tissue Eng Regen Med. 2017 May;11(5):1619-1629. doi: 10.1002/term.2079. Epub 2015 Sep 7. PMID 26876895
- [Background] Zheng C, Zhu Q, Liu X, Huang X, He C, Jiang L, Quan D, Zhou X, Zhu Z. Effect of platelet-rich plasma (PRP) concentration on proliferation, neurotrophic function and migration of Schwann cells in vitro. J Tissue Eng Regen Med. 2016 May;10(5):428-36. doi: 10.1002/term.1756. Epub 2013 May 31. PMID 23723151
- [Background] Anjayani S, Wirohadidjojo YW, Adam AM, Suwandi D, Seweng A, Amiruddin MD. Sensory improvement of leprosy peripheral neuropathy in patients treated with perineural injection of platelet-rich plasma. Int J Dermatol. 2014 Jan;53(1):109-13. doi: 10.1111/ijd.12162. Epub 2013 Oct 29. PMID 24168291
- [Background] Sanchez M, Yoshioka T, Ortega M, Delgado D, Anitua E. Ultrasound-guided platelet-rich plasma injections for the treatment of common peroneal nerve palsy associated with multiple ligament injuries of the knee. Knee Surg Sports Traumatol Arthrosc. 2014 May;22(5):1084-9. doi: 10.1007/s00167-013-2479-y. Epub 2013 Mar 22. PMID 23519544
- [Background] Raeissadat SA, Karimzadeh A, Hashemi M, Bagherzadeh L. Safety and efficacy of platelet-rich plasma in treatment of carpal tunnel syndrome; a randomized controlled trial. BMC Musculoskelet Disord. 2018 Feb 13;19(1):49. doi: 10.1186/s12891-018-1963-4. PMID 29433485
- [Background] Malahias MA, Johnson EO, Babis GC, Nikolaou VS. Single injection of platelet-rich plasma as a novel treatment of carpal tunnel syndrome. Neural Regen Res. 2015 Nov;10(11):1856-9. doi: 10.4103/1673-5374.165322. PMID 26807124
- [Background] Uzun H, Bitik O, Uzun O, Ersoy US, Aktas E. Platelet-rich plasma versus corticosteroid injections for carpal tunnel syndrome. J Plast Surg Hand Surg. 2017 Oct;51(5):301-305. doi: 10.1080/2000656X.2016.1260025. Epub 2016 Dec 6. PMID 27921443
- [Background] Wu YT, Ho TY, Chou YC, Ke MJ, Li TY, Huang GS, Chen LC. Six-month efficacy of platelet-rich plasma for carpal tunnel syndrome: A prospective randomized, single-blind controlled trial. Sci Rep. 2017 Dec;7(1):94. doi: 10.1038/s41598-017-00224-6. Epub 2017 Mar 7. PMID 28273894
- [Background] Shim JH, Ko SY, Bang MR, Jeon WJ, Cho SY, Yeom JH, Shin WJ, Kim KH, Shim JC. Ultrasound-guided greater occipital nerve block for patients with occipital headache and short term follow up. Korean J Anesthesiol. 2011 Jul;61(1):50-4. doi: 10.4097/kjae.2011.61.1.50. Epub 2011 Jul 21. PMID 21860751
- [Background] Kosinski M, Bayliss MS, Bjorner JB, Ware JE Jr, Garber WH, Batenhorst A, Cady R, Dahlof CG, Dowson A, Tepper S. A six-item short-form survey for measuring headache impact: the HIT-6. Qual Life Res. 2003 Dec;12(8):963-74. doi: 10.1023/a:1026119331193. PMID 14651415
- [Background] Nachit-Ouinekh F, Dartigues JF, Henry P, Becg JP, Chastan G, Lemaire N, El Hasnaoui A. Use of the headache impact test (HIT-6) in general practice: relationship with quality of life and severity. Eur J Neurol. 2005 Mar;12(3):189-93. doi: 10.1111/j.1468-1331.2004.00934.x. PMID 15693807
- [Background] Palamar D, Uluduz D, Saip S, Erden G, Unalan H, Akarirmak U. Ultrasound-guided greater occipital nerve block: an efficient technique in chronic refractory migraine without aura? Pain Physician. 2015 Mar-Apr;18(2):153-62. PMID 25794201
- [Background] Zipfel J, Kastler A, Tatu L, Behr J, Kechidi R, Kastler B. Ultrasound-Guided Intermediate Site Greater Occipital Nerve Infiltration: A Technical Feasibility Study. Pain Physician. 2016 Sep-Oct;19(7):E1027-34. PMID 27676673
- [Background] Gul HL, Ozon AO, Karadas O, Koc G, Inan LE. The efficacy of greater occipital nerve blockade in chronic migraine: A placebo-controlled study. Acta Neurol Scand. 2017 Aug;136(2):138-144. doi: 10.1111/ane.12716. Epub 2016 Dec 2. PMID 27910088
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Derived] Stone JE, Campbell C, Tabor JB, Bonfield S, Machan M, Shan RLP, Debert CT. Ultrasound guided platelet rich plasma injections for post-traumatic greater occipital neuralgia following concussion: a pilot randomized controlled trial. Front Neurol. 2024 Jun 7;15:1400057. doi: 10.3389/fneur.2024.1400057. eCollection 2024. PMID 38911584
- [Derived] Stone JE, Fung TS, Machan M, Campbell C, Shan RLP, Debert CT. Ultrasound-guided platelet-rich plasma injections for post-traumatic greater occipital neuralgia: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2021 Jun 22;7(1):130. doi: 10.1186/s40814-021-00867-3. PMID 34158124